CLINICAL TRIAL: NCT07375160
Title: A Retrospective, Real World Evidence (RWE) Trial Evaluating Safety and Efficacy of a Dehydrated Human Placenta Tissue (dHPT) for Wound Healing
Brief Title: Evaluating Safety and Efficacy of a Dehydrated Human Placenta Tissue (dHPT) for Wound Healing
Acronym: RETRO-PLAST
Status: Not yet recruiting | Type: Observational
Sponsor: Cellution Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: CELLBIO-2026-001
Record Dates: First submitted 2026-01-13; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Foot Ulcer (DFU); Venous Leg Ulcer (VLU); Pressure Ulcer (PU)
Keywords: Chronic Wound; Leg Wound; Amniotic; Allograft; Placenta
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer; Pressure Ulcer | interventions — Aminoimidazole Carboxamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: dHPT, AIC — Sterile dehydrated Human Amnion - Intermediate Layer - Chorion Membrane Allograft

SUMMARY:
The retrospective trial is observational, intended to stand alone, complement and integrate data collected in ongoing clinical studies to aid in establishing payor coverage in the United States (U.S.) for Cellution Biologics allograft products with real-world evidence to support the clinical adoption in patients to manage chronic or surgical wounds.

DETAILED DESCRIPTION:
Around 10.5 million Medicare beneficiaries were affected by chronic wounds in 2019. A chronic wound is generally defined as any wound that fails to heal within a reasonable timeframe. Chronic wounds can be categorized into the following four groups: arterial, pressure, diabetic, and venous. Despite the well-established standard of care for chronic wounds, which includes sharp debridement, offloading, and maintaining proper moisture balance, a notable gap remains between historical outcomes and desired results in chronic wound care.

One approach to treating chronic wounds involves the use of dehydrated human placental tissues, which are defined as 'A broad category of biomaterials, synthetic materials, or biosynthetic matrices that support repair or regeneration of injured tissues through various mechanisms of action. The application of dHTPs in chronic wound treatment provides several benefits, including creating a protective environment for healing, covering deep structures, aiding surgical closure, enhancing functional outcomes, and improving appearance. The cellular category of dHTPs includes allografts, which are human donor tissue samples intended for use in another human patient. Utilizing human amniotic membrane as an allograft displays considerable promise for chronic wound treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Wound treated with Cellution Biologics AmchoPlast, a dehydrated human placental tissue (dHPT).
* Wound present for greater than or equal to 30 days prior to treatment with dHPT.
* Wound is not infected.
* Wound surface area is greater than 1cm2 at initial assessment.
* Clinical documentation of wound treatment.

Exclusion Criteria:

* AmchoPlast dHPT product was not applied to wound.
* HbA1C >12%.
* Concurrent treatment for malignant disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be drawn from wound clinic patient population that previously received treatment of their wound with a Cellution Biologics dHPT product
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time to Closure for Target Ulcer | Up to 6 months.
  To evaluate the time to wound closure for patients treated with dHPT.

IPD SHARING:
Plan to Share IPD: No